CLINICAL TRIAL: NCT04641208
Title: Relation Between Muscle Fatigue And Time Use Of Smartphone In School Age Children
Brief Title: Time Need to Detect Mobile Phone Use to Prevent Muscle Fatigue
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: MTI University (Other)
Responsible Party: Principal Investigator, Rana Nabil Hussein Mohamed, principal investigator, MTI University
Other Study IDs: 012/002543
Record Dates: First submitted 2020-09-20; First posted 2020-11-23 (Actual); Last update posted 2020-11-23 (Actual); Status verified 2020-11

CONDITIONS: Mobile Phone Use
MeSH Terms: conditions — Cell Phone Use

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: mobile phone — The root mean square (RMS) of the signal will be calculated by using electromyography, and were normalized to the EMG data maximum voluntary isometric contraction (MVIC)

SUMMARY:
Using a smart phone while adopting a poor posture can cause various physical problems. The neck and shoulders are particularly vulnerable to pain due to smart phone use, with the muscles showing a high level of muscle fatigue, resulting in exhaustion and pain, Therefore, determining the durable time to use the smart phone will protect us from abnormal posture and protect our muscle and ligaments.

Furthermore avoid the incorrect position of use smartphone position.

DETAILED DESCRIPTION:
-Purpose of the study:

To investigate the electrical muscle activity during used mobile phone

-Back ground :

Using a smart phone while adopting a poor posture can cause various physical problems. The neck and shoulders are particularly vulnerable to pain due to smart phone use, with the muscles showing a high level of muscle fatigue, resulting in exhaustion and pain, Therefore, determining the durable time to use the smart phone will protect us from abnormal posture and protect our muscle and ligaments.

Furthermore avoid the incorrect position of use smartphone position.

-Hypotheses:

There are no statistical significant relation between time of used smart phone and muscle fatigue.

-Subjects:

One hundred fifty healthy children of both genders will participate in this study.

* Inclusion criteria:

  1. Their ages ranges from 12-14 years.
  2. Subjects of school age childhood.
  3. Not rolled on any regular athletic activity.
  4. Children should be at the same socioeconomic level.
* Exclusion criteria:

  1. Individual with neck pain
  2. Any upper limb and spinal deviation.
  3. Worker children.
* Instrumentation:

  •Surface Electromyography (EMG)
* Design of the study:

All subjects shouldn't use the phone for an hour before the measurement Each child setting in a chair with their feet on the floor and the elbow slight flexion, holding a smartphone in favorite position of used smart phone.

ELIGIBILITY:
Inclusion Criteria:

1. Their ages ranges from 12-14 years.
2. Subjects of school age childhood.
3. Not rolled on any regular athletic activity.
4. Children should be at the same socioeconomic level

Exclusion Criteria:

1. Individual with neck pain
2. Any upper limb and spinal deviation.
3. Worker children.

Ages: 12 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: All subjects shouldn't use the phone for an hour before the measurement Each child setting in a chair with their feet on the floor and the elbow slight flexion, holding a smartphone in favorite position of used smart phone using EMG surface electrode to record the muscle activity of the upper trapezius (UT), brachioradialis (BR), flexor carpi ulnaris (FCU), and abductor pollicis brevis (APB) during phone operation EMG signals are detected and the motor unite potential are measured until detecting changes in motor action potential. The root mean square (RMS) of the signal will be calculated, and were normalized to the EMG data maximum voluntary isometric contraction (MVIC)
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-02-10 (Actual); Primary Completion 2021-02-10 (Estimated); Study Completion 2021-03-10 (Estimated)

PRIMARY OUTCOMES:
Maximum voluntary contraction and Root main square | 1 day
  Maximum voluntary contraction and Root main square by using electromyography (EMG) of the upper trapezius (UT), brachioradialis (BR), flexor carpi ulnaris (FCU), and abductor pollicis brevis (APB) during phone operation

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Pysical Therapy, 6 Oct University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Statistical Analysis Plan (2019-11-12): https://cdn.clinicaltrials.gov/large-docs/08/NCT04641208/SAP_000.pdf